## Impact of Self-Awareness in Stress, Burnout, Self-Compassion and Compassion in medical students

## 096/2019

## 1 June 2020 version

- 1. I declare that I have read the form and voluntarily agree to participate in this study.
- 2. I have been informed of the nature, aims, risks, probable duration of the study, and what is expected of me.
- 3. I have had the opportunity to ask questions about the study and have understood the answers and information given to me. At any time I may ask further questions of the physician in charge of the study. During the study and whenever I want, I can receive important information that arises during the study that may change my willingness to continue to participate.
- 4. I agree that you will use information regarding my medical history and treatments with strict respect for medical confidentiality and anonymity. My data will be kept strictly confidential. I consent to consultation of my data only by persons designated by the sponsor and by representatives of regulatory authorities.
- 5. I agree to follow all instructions given to me during the study. I agree to cooperate with the doctor and inform him/her immediately of changes in my state of health and well-being and of all unexpected and unusual symptoms that occur.
- 6. I consent to the use of the results of the study for scientific purposes only and, in particular, I agree that these results may be disclosed to the appropriate health authorities.
- 7. I accept that the data generated during the study will be computerized by the sponsor or someone else designated by him/her. I may exercise my right of rectification and/or opposition.
- 8. I am aware that I am free to withdraw from the study at any time, without having to justify my decision and without compromising the quality of my medical care. I am aware that the physician has the right to decide on my premature withdrawal from the study and will inform me of the cause of such withdrawal.
- 9. I have been informed that the study may be discontinued by decision of the investigator, sponsor, or regulatory authorities.

I declare that I have read, understood and received the required information, that I am informed, and that I agree to participate voluntarily in the study.

Translated with www.DeepL.com/Translator (free version)